CLINICAL TRIAL: NCT00636792
Title: A Phase II Study of VELCADE (Bortezomib) in Combination With Bendamustine and Rituximab in Subjects With Relapsed or Refractory Follicular Lymphoma
Acronym: VERTICAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C05011
Record Dates: First submitted 2008-03-11; First posted 2008-03-14 (Estimated); Results first posted 2011-06-22 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Bortezomib; Bendamustine Hydrochloride; Rituximab

ARMS (1):
- 1 (Experimental): This is a phase 2, single-arm, open label, multicenter study evaluating the efficacy and safety of the combination of VELCADE, bendamustine, and rituximab in subjects with relapsed or refractory follicular lymphoma, who have received 4 or more doses of rituximab. Subjects may be sensitive or refractory to prior therapies, including rituximab.
  Interventions: Drug: VELCADE; Drug: Bendamustine; Drug: Rituximab

INTERVENTIONS:
Drug: VELCADE — VELCADE administered as a 3- to 5-second intravenous (IV) bolus prior to Bendamustine and Rituximab on Days 1,8,15 and 22 of each cycle.
Drug: Bendamustine — Bendamustine administered IV over 30-60 minutes after VELCADE on Days 1 and 2 of each cycle
Drug: Rituximab — Rituximab administered by IV infusion after VELCADE and Bendamustine on Days 1, 8, 15 and 22 of Cycle 1, and on Day 1 of Cycles 2, 3, 4 and 5

SUMMARY:
This is a phase 2, single-arm, open label, multicenter study evaluating the efficacy and safety of the combination of VELCADE, bendamustine, and rituximab in subjects with relapsed or refractory follicular lymphoma, who have received 4 or more doses of rituximab. Subjects may be sensitive or refractory to prior therapies, including rituximab.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject 18 years of age or older
* Pathological diagnosis of follicular lymphoma (any grade)
* Documented relapse or progression following prior antineoplastic therapy
* Have received 4 or more prior doses of rituximab
* At least 1 measurable tumor mass (>1.5 cm in the long axis and >1.0 cm in the short axis that has not been previously irradiated, or has grown since previous irradiation
* No clinically significant central nervous system lymphoma
* Karnofsky performance status (KPS) ≥50 (equivalent to Eastern Cooperative Group Oncology Group [ECOG] status ≤2

Exclusion Criteria:

* Diagnosed or treated for a malignancy other than non-Hodgkin's lymphoma (NHL) within 2 years of first dose, or who were previously diagnosed with a malignancy other than NHL and have any radiographic or biochemical marker evidence of malignancy. Subjects with prostate cancer who were treated with definitive radiotherapy and have a serum prostate-specific antigen (PSA) <1 ng/mL are not excluded. Subjects are also not excluded if they have had basal cell or squamous cell carcinoma of the skin that was completely resected, or any in situ malignancy that was adequately treated.
* Prior treatment with VELCADE® or bendamustine
* Antineoplastic (including unconjugated therapeutic antibodies and toxin immunoconjugates), experimental, or radiation therapy within 3 weeks before Day 1 of Cycle 1
* Nitrosoureas within 6 weeks before Day 1 of Cycle 1
* Radioimmunoconjugates within 10 weeks before Day 1 of Cycle 1
* Autologous stem cell transplant within 3 months before Day 1 of Cycle 1, or prior allogeneic stem cell transplant at any time
* Major surgery within 2 weeks before Day 1 of Cycle 1
* Platelet transfusion within 7 days of Day 1 of Cycle 1 (applies to subjects enrolled in the dose escalation phase only. This does not apply to subjects enrolled in phase 2 of the study).
* Ongoing therapy with corticosteroids. Prednisone ≤15 mg per day or its equivalent is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2008-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (2):
- United States (2):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - MidDakota Clinic - Cancer Treatment and Research Center, Bismarck, North Dakota

RESULTS

PARTICIPANT FLOW:
Groups:
- VELCADE, Bendamustine, Rituximab (VBR) Treatment: Patients receive bortezomib 1.6 mg/m^2 IV on days 1, 8, 15, and 22 of each 35-day cycle; bendamustine 50-90 mg/m^2 IV on days 1 and 2 of each cycle; rituximab 375 mg/m^2 IV on days 1, 8, 15 and 22 of cycle 1 and on day1 of cycles 2, 3, 4, and 5. Total treatment duration is 5 cycles.
Period: Overall Study
Arm/Group | VELCADE, Bendamustine, Rituximab (VBR) Treatment
Started | 73
Completed | 40
Not Completed | 33
Not completed — Adverse Event | 16
Not completed — Physician Decision | 7
Not completed — Progressive Disease | 4
Not completed — Withdrawal by Subject | 3
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Arm/Group | VELCADE, Bendamustine, Rituximab (VBR) Treatment
Number analyzed (Participants) | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 49
  >=65 years | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 59.8 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 44
Region of Enrollment [Number; unit: participants]
  United States | 73

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response
Description: Response is assessed by investigator according to International Working Group (IWG) criteria. Complete response requires disappearance of all evidence of disease.
Time Frame: 12 weeks after the last subject completes their end of treatment visit.
Population: Response-evaluable population is defined at patients treated with 90 mg/m^2 bendamustine, received at least one dose of any study drug, and had at least one post baseline response assessment.
Measure: Number; unit: participants
Arm/Group | VELCADE, Bendamustine, Rituximab (VBR) Treatment
Number analyzed (Participants) | 60
participants | 32

2. Secondary Outcome: Number of Participants With Overall Response (Complete and Partial Response)
Description: Response is assessed by investigator according to International Working Group (IWG) criteria. Complete response requires disappearance of all evidence of disease. Partial response requires regression of measurable disease and no new sites.
Time Frame: 12 weeks after the last subject completes their end of treatment visit
Measure: Number; unit: participants
Arm/Group | VELCADE, Bendamustine, Rituximab (VBR) Treatment
Number analyzed (Participants) | 60
participants | 53

ADVERSE EVENTS:
Time Frame: Start from first dose of any study drug, end at 30 days post last dose of any study drug, or start of subsequent antineoplastic therapy, whichever occurs first.
Arm/Group | VELCADE, Bendamustine, Rituximab (VBR) Treatment
Serious Adverse Events (participants affected / at risk) | 25/73
Other Adverse Events (participants affected / at risk) | 72/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VELCADE, Bendamustine, Rituximab (VBR) Treatment (N=73)
Pneumonia NOS (Infections and infestations) | 2
Bronchitis NOS (Infections and infestations) | 1
Pulmonary mycosis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Urinary tract infection NOS (Infections and infestations) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Pancytopenia (Blood and lymphatic system disorders) | 1
Leukopenia NOS (Blood and lymphatic system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhoea NOS (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Vomiting NOS (Gastrointestinal disorders) | 2
Ileus paralytic (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 3
Fatigue (General disorders) | 1
Weakness (General disorders) | 1
Disease progression NOS (General disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Syncope (Nervous system disorders) | 1
Peripheral neuropathy NOS (Nervous system disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 1
Cholecystitis acute NOS (Hepatobiliary disorders) | 1
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 1
Tumour lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Orthostatic hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VELCADE, Bendamustine, Rituximab (VBR) Treatment (N=73)
Constipation (Gastrointestinal disorders) | 33
Abdominal pain NOS (Gastrointestinal disorders) | 13
Abdominal pain upper (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 9
Mouth ulceration (Gastrointestinal disorders) | 4
Pharyngolaryngeal pain (Gastrointestinal disorders) | 6
Flatulence (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 5
Rigors (General disorders) | 27
Chest pain (General disorders) | 4
Oedema lower limb (General disorders) | 7
Dizziness (excl vertigo) (Nervous system disorders) | 17
Dysgeusia (Nervous system disorders) | 5
Headache NOS (Nervous system disorders) | 20
Peripheral sensory neuropathy (Nervous system disorders) | 10
Hypoaesthesia (Nervous system disorders) | 4
Anaemia NOS (Blood and lymphatic system disorders) | 26
Neutropenia (Blood and lymphatic system disorders) | 25
Lymphopenia (Blood and lymphatic system disorders) | 4
Pruritus NOS (Skin and subcutaneous tissue disorders) | 6
Rash NOS (Skin and subcutaneous tissue disorders) | 6
Night sweats (Skin and subcutaneous tissue disorders) | 5
Skin lesion NOS (Skin and subcutaneous tissue disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 17
Appetite decreased NOS (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 14
Hypomagnesaemia (Metabolism and nutrition disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 10
Pain in limb (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Upper respiratory tract infection NOS (Infections and infestations) | 6
Herpes simplex (Infections and infestations) | 7
Oral candidiasis (Infections and infestations) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Rhinitis allergic NOS (Respiratory, thoracic and mediastinal disorders) | 4
Insomnia (Psychiatric disorders) | 16
Anxiety NEC (Psychiatric disorders) | 9
Depression NOS (Psychiatric disorders) | 8
Hypotension NOS (Vascular disorders) | 7
Phlebitis NOS (Vascular disorders) | 4
Hypertension NOS (Vascular disorders) | 4
Vision blurred (Eye disorders) | 5
Eye irritation (Eye disorders) | 4
Urinary frequency (Renal and urinary disorders) | 4
Dysuria (Renal and urinary disorders) | 4
Palpitations (Cardiac disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No